CLINICAL TRIAL: NCT07094802
Title: Comparison of Intrathecal Bupivacaine With and Without Morphine for Post-operative Analgesia in Parturients Undergoing Elective Cesarean Section: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Megha Patrabansha, Dr., Resident, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IT Morphine CS -072114
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pain; Cesarean Delivery; Analgesia, Obstetrical
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine; Morphine; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morphine Group (Active Comparator): This group will receive 2.2 ml of 0.5% hyperbaric bupivacaine + 100 mcg (0.1 ml of 1 mg/ml) Morphine intrathecally during spinal anesthesia
  Interventions: Drug: Intrathecal morphine with bupivacaine
- Bupivacaine Group (Placebo Comparator): This group will receive 2.2 ml of 0.5% hyperbaric bupivacaine during spinal anesthesia
  Interventions: Drug: Hyperbaric Bupivicaine

INTERVENTIONS:
Drug: Intrathecal morphine with bupivacaine — Participants will receive 100 mcg intrathecal morphine along with 2.2ml of 0.5% hyperbaric bupivacaine
  Other Names: morphine; opioids; intrathecal morphine
  Arms: Morphine Group
Drug: Hyperbaric Bupivicaine — 0.5% hyperbaric Bupivacaine 2.2 ml
  Other Names: Bupivacaine; hyperbaric bupivacaine
  Arms: Bupivacaine Group

SUMMARY:
The goal of this clinical trial is to compare intrathecal bupivacaine with or without morphine for postoperative analgesia in patients undergoing elective cesarean section. The main questions it aims to answer are:

Is intrathecal bupivacaine with morphine superior to intrathecal bupivacaine alone for postoperative analgesia for parturients undergoing cesarean section? What is the duration of analgesia in the two groups? Researchers will compare drug intrathecal bupivacaine with morphine to a iintrathecal bupivacaine alone to see if intrathecal morphine has benefits for psotoperative analgesia .

Participants will:

Get intrathecal bupivacaine with Morphine or intrathecal bupivacaine alone during spinal anesthesia for cesarean section.

They will be followed up for NRS pain scores and side effects for 24 hours. Time to need of first rescue analgesic will be noted

ELIGIBILITY:
Inclusion Criteria:

* Parturients undergoing elective caesarean section under Spinal anesthesia
* ASA PS II, III
* > 18 years

Exclusion Criteria:

* Refusal to Participate
* Contraindications to spinal anaesthesia and adjuvants INR ≥ 1.5 Plateletes < 1,00,000/cumm Severe aortic stenosis, and/or severe mitral stenosis Infection at lumbar puncture site Known allergy to local anesthetics and opioids
* Communication barrier
* Height <150 cm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 92 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Time to need of first rescue analgesic | within 24 hours
  time of spinal anesthesia to time of demand of first rescue analgesic
NRS score | 24 hours
  comapre NRS score at 0,1,6,12,18,24 hours between the groups

SECONDARY OUTCOMES:
24 hours analgesic consumption | 24 hours
  consumtion of total analgesic in first 24 hours